CLINICAL TRIAL: NCT00775788
Title: Autologous Fat Grafting to the Breast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Kamran Khoobehi MD FACS, LSUHSC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7006
Record Dates: First submitted 2008-10-15; First posted 2008-10-20 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-10

CONDITIONS: Micromastia; Breast Ptosis; Implant Failure; Breast Reconstruction; Congenital Malformations
Keywords: Fat Injection to Breast; Fat Grafting to Breast
MeSH Terms: conditions — Congenital Abnormalities | interventions — Mammaplasty; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Implant Failure (Experimental)
  Interventions: Procedure: Autologous Fat Grafting to Breasts
- Post mastectomy breast reconstruction (Experimental)
  Interventions: Procedure: Autologous Fat Grafting to Breasts
- Congenital malformations (Experimental)
  Interventions: Procedure: Autologous Fat Grafting to Breasts
- Breast Ptosis (Experimental)
  Interventions: Procedure: Autologous Fat Grafting to Breasts
- Micromastia (Experimental)
  Interventions: Procedure: Autologous Fat Grafting to Breasts
- Asymmetric Breasts (Experimental)
  Interventions: Procedure: Autologous Fat Grafting to Breasts

INTERVENTIONS:
Procedure: Autologous Fat Grafting to Breasts — Fat injection of Fat to breasts
  Other Names: Breast Reconstruction; Implant related complications; Mastectomy

SUMMARY:
Structural fat grafting is a form of tissue transfer where the autologous fat is harvested and subsequently transferred to a different region of the body at the same setting. It is an excellent technique for filling soft tissue and contour defects. Fat has the benefit of being abundantly available and easy to harvest. Further more, it is cheap and autogenous and thus lacks the side effects of synthetic fillers or implants. Autogenous fat transfer is a relatively common procedure performed by plastic and reconstructive surgeons. The goal of fat grafting is to provide the patient with a predictable, long lasting autogenous soft tissue augmentation. Autogenous fat transfer has been used extensively as an adjunct to facial rejuvenation. As well it has been applied to body contouring and augmentation of the hips, trochanteric areas, thighs and buttocks, back, torso and breast. The transfer of autologous fat dates back to 1890s and more specifically as injectable grafts since the 1920s. However, over the past 20 years the popularity of structural fat grafting has increased as a contouring modality. Fat transfer to the breast, popularized by Coleman, has been performed internationally since the 1990s. Despite the duration, the literature lacks accurate outcomes data on fat transfer to the breast and questions regarding the viability of adipocytes after the transfer exist. Sources from various publications show cell viability of up to 100% however studies of long term clinical outcomes quote rates of 10% to 80%.

DETAILED DESCRIPTION:
Our goal with this study is to prospectively acquire information with our protocol that will outline the accurate long-term outcomes of fat transfer to the breast. Currently, fat grafting to the breast is a treatment option in conditions such as micromastia, breast ptosis, post mastectomy breast reconstruction, asymmetric breasts, congenital malformations of breast development and for treatment of complications associated with implant augmentation mammoplasty. In addition to fat grafting, the current surgical treatment for these conditions is mainly based on techniques requiring implant augmentation or reconstruction. Although the safety of saline implants has been well studied and documented, this data cannot be extrapolated for the newer generation silicone implants and other alternatives such as fat grafting need to be investigated. Also implant augmentation and reconstruction comes at the price of capsular contracture, implant deflation, infection and more future corrective surgeries. We plan to prospectively study the outcomes of fat grafting in patients with these conditions for a period of 5 years. The collected information will be entered into a database and will be prospectively collected and reviewed. Patients demographics, information obtained during the preoperative and postoperative visits along with the pertinent findings regarding the fat transfer to the breast will be collected into the database for our investigation.

ELIGIBILITY:
Inclusion Criteria:

* Women with the following conditions micromastia, breast ptosis, post mastectomy breast reconstruction, asymmetric breasts, congenital malformations of breast development and for treatment of complications associated with implant augmentation mammoplasty.

Exclusion Criteria:

* A volunteer who has a positive pregnancy test
* A volunteer who has had a cardiac stent placed within the last two months
* A volunteer with a known, current substance abuse
* A volunteer with a bleeding diathesis
* Untreated breast cancer
* A volunteer who smokes cigarettes
* Medical Conditions including untreated hypertension, renal disease, diabetes mellitus

Ages: 17 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
3 Dimensional volumetric analysis of results and photographic analysis by board certified plastic surgeons. | 3 months, 6 months and annually

SECONDARY OUTCOMES:
Patient satisfaction with cosmetic and reconstructive results | 3 months, 6 months and annually

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Khoobehi, MD, Principal Investigator — LSUHSC; Alireza Sadeghi, MD, Study Director — LSUHSC
Locations (2):
- United States (2):
  - Houma Outpatient Surgery Center, Metairie, Louisiana
  - Medical Center of Louisiana New Orleans, LSU Health Sciences Center, New Orleans, Louisiana

REFERENCES:
- [Result] Coleman SR, Saboeiro AP. Fat grafting to the breast revisited: safety and efficacy. Plast Reconstr Surg. 2007 Mar;119(3):775-85; discussion 786-7. doi: 10.1097/01.prs.0000252001.59162.c9. PMID 17312477
- See also: Related Info — http://www.khoobehi.com